CLINICAL TRIAL: NCT04805710
Title: The Efficacy and Safety of Clopidogrel Combined With Rivaroxaban and Aspirin in Patients With Coronary Heart Disease and Gastrointestinal Diseases Undergoing PCI：a Randomized Controlled Study
Brief Title: Rivaroxaban or Aspirin in Patients With CHD & GD Undergoing PCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, Director of cardiology, Shenyang Northern Hospital, Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShenyangNH
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Rivaroxaban
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clopidogrel combined with aspirin arm (No Intervention): Patients selected in the clopidogrel combined with aspirin arm will receive clopidogrel 75 mg once daily and aspirin 100 mg once daily.
- clopidogrel combined with rivaroxaban arm (Experimental): Patients selected in the clopidogrel combined with rivaroxaban arm will receive clopidogrel 75 mg once daily and rivaroxaban 10 mg once daily.
  Interventions: Drug: clopidogrel combined with rivaroxaban arm

INTERVENTIONS:
Drug: clopidogrel combined with rivaroxaban arm — Patients who have been selected will be randomized to the clopidogrel combined with rivaroxaban arm. clopidogrel 75 mg once daily and rivaroxaban 10 mg once daily
  Other Names: clopidogrel combined with rivaroxaban
  Arms: clopidogrel combined with rivaroxaban arm

SUMMARY:
The aim of this study is to assess the efficacy and safety of rivaroxaban or aspirin combined with clopidogrel in patients with coronary heart disease and gastrointestinal diseases undergoing PCI.

DETAILED DESCRIPTION:
Background：Aspirin combined with P2Y12 receptor antagonist are the antithrombotic basis of percutaneous coronary intervention (PCI) for coronary heart disease. Guidelines at home and abroad recommend that patients with stable coronary heart disease need double antiplatelet therapy for 6 months, and patients with acute coronary syndrome need double antiplatelet therapy for 12 months to prevent stent thrombosis and reduce the risk of ischemic or atherosclerotic thrombosis events, including stent thrombosis, recurrent myocardial infarction and cardiogenic death. Aspirin can inhibit the activity of cyclooxygenase in gastrointestinal tract, causing gastrointestinal mucosal epithelial injury and bleeding. For patients with gastrointestinal diseases, the risk of bleeding is higher after taking aspirin for a long time. 48.7% of PCI patients suffered from bleeding in digestive tract, so it is very important to protect gastrointestinal mucosa. In the past, patients with coronary heart disease who were accompanied by gastrointestinal diseases and could not tolerate aspirin often delayed PCI or conservative treatment with drugs, and the prognosis was very poor. In the study of patients with coronary heart disease complicated with atrial fibrillation undergoing PCI, it is concluded that the bleeding rate in the clopidogrel combined with rivaroxaban group is lower and the curative effect is not inferior to that of triple antithrombotic regimen. Whether rivaroxaban can replace aspirin for coronary heart disease complicated with gastrointestinal diseases has no research evidence and no relevant guidelines.

Methods:Patients who have been selected will be randomized to the clopidogrel combined with rivaroxaban arm versus the clopidogrel combined with aspirin arm. Patients selected in the clopidogrel combined with rivaroxaban arm will receive clopidogrel 75 mg once daily and rivaroxaban 10 mg once daily. Patients selected in the clopidogrel combined with aspirin arm will receive clopidogrel 75 mg once daily and aspirin 100 mg once daily. The therapy will last for at least six months in the both arms. The primary endpoints will be evaluated at six-months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged from 18 to 75 years
* Patient presents with Non-ST-segment elevation acute coronary syndrome (NSTEMI) combined with GRACE score < 140 points or stable coronary artery disease (SCAD)
* Patient has gastrointestinal diseases (Gastrointestinal diseases are defined as acute or chronic gastritis, erosive gastritis, gastrointestinal bleeding or peptic ulcer healing for 1-12 months, gastrointestinal dysfunction diagnosed by a specialist, and gastrointestinal tumor to be operated on)
* Patient with gastrointestinal bleeding or ulcer in the past one year ago has stomach pain, abdominal distension or other discomfort after taking aspirin, but they can tolerate it
* Patient voluntarily signs informed consent form

Exclusion Criteria:

* Patient presents with Non-ST-segment elevation acute coronary syndrome (NSTEMI) combined with GRACE score >140 points or ST-segment elevation acute myocardial infarction (STEMI)
* Patient with intracranial hemorrhage (within one month) or bleeding of important organs or other than recent surgery for gastrointestinal tumors
* Platelet count <100 000/μL
* Hemoglobin <100g/L
* Patient with active liver diseases or ALT >3 × the upper limit of the normal range or AST>3 × the upper limit of the normal range
* Patient with severe renal insufficiency (eGFR <30ml/min/1.73m2 based on simplified MDRD equation or CrCl <30ml/min based on Cockcroft-Gault equation)
* Patient with active stage of digestive tract ulcer
* Patient with less weight （Weight less than 45kg）
* Allergic to aspirin or rivaroxaban
* Patient has no intention of PCI treatment
* Patient has a malignancy or a life expectancy of less than six months
* Patient is pregnant, breastfeeding, or planning to become pregnant within 6 months
* Patient should take potent CYP3A4 inhibitors and p-gp inhibitors for a long time(such as Ketoconazole, voriconazole, nefazodone, erythromycin)
* Patient should take medium and strong CYP2C19 inhibitors (such as omeprazole, esomeprazole, fluconazole, etc.) or CYP2C19 inducers (such as rifampicin) which are known to interact with clopidogrel for a long time
* Patient is not expected to tolerate six months of medication
* No informed consent can be obtained or any situation that the researcher thinks is not suitable for participating in this study
* Patient is participating in other ongoing clinical studies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1020 (Estimated)
Dates: Start 2021-03-17 (Estimated); Primary Completion 2022-09-16 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of moderate and serve bleeding events which is identified by Bleeding Academic Research Consortium (BARC) | 6 months
  Bleeding Academic Research Consortium (BARC)

SECONDARY OUTCOMES:
Occurrence of main adverse cardiovascular and cerebrovascular events (MACCE) | 6 months
  MACCE will include all-cause death, non-fatal stroke, non-fatal myocardial infarction (MI) and ischemia driven revascularization.